CLINICAL TRIAL: NCT00978835
Title: Tailored Case Management for Diabetes and Hypertension
Acronym: TEACH-DM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00002325; 1R01DK074672 (NIH)
Record Dates: First submitted 2009-09-15; First posted 2009-09-17 (Estimated); Last update posted 2014-07-15 (Estimated); Status verified 2014-07

CONDITIONS: Diabetes; Hypertension
Keywords: Diabetes; Hypertension; Physical Activity; Diet; Medication Adherence
MeSH Terms: conditions — Diabetes Mellitus; Hypertension; Motor Activity; Medication Adherence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nurse case management (Experimental): Telephone calls by a nurse every two months to assess adherence to diet, physical activity, and pill-taking regimens. The nurse will then identify barriers to adherence to these recommendations and use motivational interviewing approaches to offer solutions to the barriers identified. No changes to medication are made.
  Interventions: Behavioral: Tailored telephone-based case management
- Nurse Education (Active Comparator): Didactic, non-interactive education by a nurse on general health topics.
  Interventions: Behavioral: Nurse Education

INTERVENTIONS:
Behavioral: Tailored telephone-based case management — Telephone calls by a nurse every two months to assess adherence to diet, physical activity, and pill-taking regimens. The nurse will then identify barriers to adherence to these recommendations and use motivational interviewing approaches to offer solutions to the barriers identified. No changes to medication are made.
  Arms: Nurse case management
Behavioral: Nurse Education — Didactic, non-interactive education by a nurse on general health topics. Calls are made every two months.
  Arms: Nurse Education

SUMMARY:
Diabetes and hypertension co-exist in approximately 10 million people in the USA and constitute severe risk factors for the development of such complications as heart and kidney disease. The investigators propose a randomized controlled trial in patients of community primary care practices to study a tailored telephone-administered behavioral intervention to improve control of blood pressure and blood sugar in patients with both hypertension and diabetes. The investigators hypothesize that 20% more patients talking to a nurse every other month about ways to improve blood pressure and blood sugar control will bring their blood pressure under control when compared to patients who talk with the nurse only about general health issues. If successful in improving control of these diseases this intervention can easily be adopted in other community primary care practices to lessen the burden of diabetes and hypertension in the USA.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled and receiving primary care at one of 9 participating clinics in North Carolina
* Diagnosis of diabetes as determined by billing data
* Taking medication for diabetes
* Diagnosis of hypertension as determined by billing data
* Taking medication for hypertension
* Most recent (within one year) Hemoglobin A1c >= 7.5%

Exclusion Criteria:

* Active psychosis
* Hospitalization for stroke, myocardial infarction (MI), or coronary artery revascularization in the past 6 months
* Type I diabetes
* Does not speak English
* No access to a telephone
* Institution-dwelling or receiving comprehensive professional home health care
* Hearing or speech inadequate for long interactive phone conversations
* Terminal illness or active treatment for cancer
* Cognitive impairment too severe to understand instructions

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 377 (Actual)
Dates: Start 2008-05; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Blood Pressure | 2 years

SECONDARY OUTCOMES:
Hemoglobin A1c | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States